CLINICAL TRIAL: NCT04439760
Title: Efficacy of Superior Cervical Ganglion (SCG) Block on the Incidence and Severity of Vasospasm After Middle Cerebral Artery (MCA)Aneurysmal Surgery Using Transcranial Doppler(TCD). A Randomized Controlled Trial.
Brief Title: Superior Cervical Ganglion Block, Transcranial Doppler
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatma Ibrahim El Sayed Salman (Other)
Responsible Party: Sponsor-Investigator, Fatma Ibrahim El Sayed Salman, anesthesia assistant lecturer, Kasr El Aini Hospital
Organization: Kasr El Aini Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: transcranial Doppler
Record Dates: First submitted 2020-06-13; First posted 2020-06-19 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Brain Aneurysm; Aneurysm, Ruptured
Keywords: middle cerebral artery
MeSH Terms: conditions — Intracranial Aneurysm; Aneurysm, Ruptured

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control study. (No Intervention): No intervention
- superior cervical block. (Active Comparator): Under X-ray guidance, a 23-gauge radiofrequency top-pole needle with an active tip of 5 mm is inserted for test blockade. The needle is directed at the facet joint of the 3rd and 4th cervical vertebrae.The needle is introduced parallel to the radiographic projection and is projected as a dot approximately 1 cm anterior to the spine. The radiographic projection is then changed to lateral, and the needle is slowly advanced until the tip was situated at the anterior border of the third cervical vertebra. On the anteroposterior projection, the tip of the needle is projected over the lateral part of the facetal column. When the tip of the needle is in position, 0.3 mL of Omnipaque is injected. On the transverse projection, the contrast is distinctly anterior to anterior border of the vertebral bodies, and in the anteroposterior projection, the contrast is seen spreading in a space overlying the facetal column in a cranial as well as caudal direction.
  Interventions: Procedure: Superior Cervical Ganglion Block

INTERVENTIONS:
Procedure: Superior Cervical Ganglion Block — Under X-ray guidance, a 23-gauge radiofrequency top-pole needle with an active tip of 5 mm is inserted for test blockade. The needle is directed at the facet joint of the 3rd and 4th cervical vertebrae.The needle is introduced parallel to the radiographic projection and is projected as a dot approximately 1 cm anterior to the spine. The radiographic projection is then changed to lateral, and the needle is slowly advanced until the tip was situated at the anterior border of the third cervical vertebra. On the anteroposterior projection, the tip of the needle is projected over the lateral part of the facetal column. When the tip of the needle is in position, 0.3 mL of Omnipaque is injected. On the transverse projection, the contrast is distinctly anterior to anterior border of the vertebral bodies, and in the anteroposterior projection, the contrast is seen spreading in a space overlying the facetal column in a cranial as well as caudal direction.
  Arms: superior cervical block.

SUMMARY:
The aim of this study is to assess blood flow velocity in middle cerebral artery measured by transcranial doppler to determine the efficacy of SCG block in decreasing incidence or severity of vasospasm after MCA aneurysm surgery.

DETAILED DESCRIPTION:
Sympathetic innervation to the face and head is by superior cervical ganglion(SCG), which is the most cranial part of the sympathetic chain. It is suited in a plication of the prevertebral fascia anterior to the longuscapitis muscle and dorsal to the internal carotid artery, posteromedial to the vagus nerve at c3 level. It's mainly located at the level of the transverse processes of the second and third cervical vertebrae. However, it may reach caudally to the upper border of the fourth cervical vertebra.

Noradrenergic sympathetic nerve fibers mainly originating in the superior cervical ganglion, accompanying the carotid artery supply cerebral vasculature particularly the pial vessels.

Superior cervical ganglion block was previously tried in managing neuropathic pain, neuropathic pain in head and face region was investigated in patients using ganglionic local opioid analgesia (GLOA) at the superior cervical ganglion (SCG) ,The short-term analgesic effect of the first blockade by GLOA was significant with a mean pain reduction of 52% (p < 0.001).

Superior cervical ganglion block also used as an alternative treatment to tinnitus not responding to conventional therapy, it increases cholear blood flow and this can explain the efficacy of block.

Superior cervical ganglion block was used to improve cerebral perfusion in patients with cerebral vasospasm after aSAH.

Aneurysmal subarachnoid hemorrhage (aSAH) may develop vasospasm in 70% of patients. Morphological changes occur in the cerebral vessels after SAH, and the inflammatory response and local chemical agents are responsible for the induction of vasospasm.

Vasospasm is rare in the first 3 days after SAH, it reaches peak incidence at 7 to10 days and usually resolves by 10 to14 days after SAH.

The sympathetic system also has a role in the pathogenesis of this process, cervical sympathetic stimulation leads to constriction in intracerebral vessels and dilation occurs when these fibers are interrupted. Efflux and reuptake of the neurotransmitter may be prevented by sympathectomy.

Common treatments to reduce vasospasm include ;triple H therapy (hypertension ,hypervolemia and hemodilution), intraarterial infusion of Smooth muscle relaxants (papaverine, Verapamil) and endovascular balloon angioplasty . Also (nimodipine) calcium channel blocker administration is used as a prophylactic measures.

Transcranial doppler (TCD) is a non-invasive technique which can be used to observe velocity, direction and properties of blood flow in the cerebral arteries by means of a pulsed ultrasonic beam, based on the Doppler effect of ultrasounds concerning frequency variations in sound waves as a result of relative motion between source and signal receiver. It was previously used in traumatic brain injury(TBI),stroke, anesthesia and intensive care.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 18 to 70 years.
* Genders eligible for study: both sexes.
* ASA I-II.
* GCS (13-15)

Exclusion Criteria:

* Patient refusal
* Contraindications to regional anesthesia (Bleeding disorders, Use of any anti-coagulants, local infection).
* Known allergy to local anesthetics.
* ASA III-IV.
* Patients aged less than 18 or more than 70.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline Blood flow velocity in middle cerebral artery measured by transcranial doppler (TCD) | The day before surgery (TCD0), Postoperative at day 3 and day 7 (TCD3 & TCD7)
  Change in Blood flow velocity in patients with ruptured aneurysmal subarachnoid hemorrhage undergoing MCA aneurysmal surgeries measured by transcranial doppler

SECONDARY OUTCOMES:
Incidence or severity of MCA postoperative spasm over 14 days. | within 14 days
  TCD MCA vasospasm diagnostic criteria :
  Proximal MCA vasospasm can be diagnosed by any of the following:
  MCA Mean flow velocities of > 200 cm/s, Rapid rise in flow velocities (> 65 cm/s in one day), or Lindegaard ratio (VMCA/VICA >6).
Change from baseline heart rate | Baseline (Before surgery) ,after induction the block and at the end of surgery
  Heart rate will be measured
Change from baseline mean arterial blood pressure | Baseline (Before surgery) ,after induction the block and at the end of surgery
  Mean arterial blood pressure will be measured
Change from baseline oxygen saturation (Sao2) | Baseline (Before surgery) ,after induction the block and at the end of surgery
  Oxygen saturation (Sao2) will be measured
Incidence of complications (Nerve injury, Hematoma formation, LA toxicity, Sensory or motor deficit, respiratory depression). | within 14 days
  Incidence of complications (Nerve injury, Hematoma formation, LA toxicity, Sensory or motor deficit, respiratory depression) will be assisted
Glasgow coma scale | Baseline (Preopetative), at day 3 and day 7
  Glasgow coma scale will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Salman, Master, Principal Investigator — Kasr El Aini Hospital
Locations (1):
- kasr Al Ainy hospital, Cairo, Egypt

REFERENCES:
- [Background] Siegenthaler A, Haug M, Eichenberger U, Suter MR, Moriggl B. Block of the superior cervical ganglion, description of a novel ultrasound-guided technique in human cadavers. Pain Med. 2013 May;14(5):646-9. doi: 10.1111/pme.12061. Epub 2013 Feb 25. PMID 23438374
- [Background] Tuor UI. Local distribution of the effects of sympathetic stimulation on cerebral blood flow in the rat. Brain Res. 1990 Oct 8;529(1-2):224-31. doi: 10.1016/0006-8993(90)90831-u. PMID 2282493
- [Background] Kurth CD, Wagerle LC, Delivoria-Papadopoulos M. Sympathetic regulation of cerebral blood flow during seizures in newborn lambs. Am J Physiol. 1988 Sep;255(3 Pt 2):H563-8. doi: 10.1152/ajpheart.1988.255.3.H563. PMID 3137827
- [Background] Koning HM, Dyrbye BA, van Hemert FJ. Percutaneous Radiofrequency Lesion of the Superior Cervical Sympathetic Ganglion in Patients with Tinnitus. Pain Pract. 2016 Nov;16(8):994-1000. doi: 10.1111/papr.12348. Epub 2015 Aug 27. PMID 26311111
- [Background] Rumalla K, Smith KA, Arnold PM, Mittal MK. Subarachnoid Hemorrhage and Readmissions: National Rates, Causes, Risk Factors, and Outcomes in 16,001 Hospitalized Patients. World Neurosurg. 2018 Feb;110:e100-e111. doi: 10.1016/j.wneu.2017.10.089. Epub 2017 Oct 26. PMID 29107164
- [Background] Sharma AK, Bathala L, Batra A, Mehndiratta MM, Sharma VK. Transcranial Doppler: Techniques and advanced applications: Part 2. Ann Indian Acad Neurol. 2016 Jan-Mar;19(1):102-7. doi: 10.4103/0972-2327.173407. PMID 27011639